CLINICAL TRIAL: NCT02496156
Title: Shared Medical Decision Making in Pediatric Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nemours Children's Clinic (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: PCORI 805
Record Dates: First submitted 2015-04-23; First posted 2015-07-14 (Estimated); Results first posted 2024-02-01 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2023-05

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: type 1 diabetes mellitus; adolescence; adherence; insulin pump; continuous subcutaneous insulin infusion; continuous glucose monitor; shared medical decision making
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: 2 group (Usual Clinical Practice or Shared Medical Decision Making X 5 time points (0, 3, 6, 9 and 12 months) repeated measures randomized treatments design.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Clinical Practice (UCP) (Active Comparator): UCP participants will receive the same clinical and educational management for candidates for insulin pump or continuous glucose monitoring that is received by similar patients who are not enrolled in this study. The respective endocrinology practices at the enrolling sites all strive to meet or exceed the current American Diabetes Association Standards for Clinical Practice in the management of type 1 diabetes in this population. Thorough patient education is the cornerstone of that care, especially regarding the incorporation of insulin pumps and continuous glucose monitors into the treatment regimen for a given patient.
  Interventions: Behavioral: Usual Clinical Practice
- Shared Medical Decision Making (SMDM) (Experimental): Participants randomized to SMDM receive all components of UCP supplemented with access to the decision aid website pertinent to the medical decision of interest (pump or CGM). Adolescents and parents will receive password-protected, secure access to the decision for their use until a decision is reached. The platform will then generate a summary report that the adolescent and parent will discuss with a diabetes nurse and then a visit with the treating endocrinologist will be scheduled to conclude the SMDM intervention for that adolescent and parent.
  Interventions: Behavioral: Shared Medical Decision Making

INTERVENTIONS:
Behavioral: Usual Clinical Practice — Diabetes management and education related to insulin pump or continuous glucose monitor as currently practiced at the enrolling site.
  Arms: Usual Clinical Practice (UCP)
Behavioral: Shared Medical Decision Making — Access to and use of multimedia decision aid websites to facilitate adolescent and parent decision making about incorporating these devices into the diabetes management regimen.
  Arms: Shared Medical Decision Making (SMDM)

SUMMARY:
This work is testing a shared medical decision making intervention for adolescents with type 1 diabetes and their parents who are candidates for adding either an insulin pump or continuous glucose monitor to their treatment plan. The first half of the work consisted of the stakeholder driven design, construction and refinement of web-delivered multimedia decision aids for each of these decisions. The randomized controlled trial of that intervention began enroling participants in February 2015. A sample of 166 eligible adolescents who receive care at an operating entity of the Nemours Children's Health System will be enrolled and randomized to either Usual Clinical Practice alone or augmented by the Shared Medical Decision Making intervention. Primary outcomes include measures of engagement with the pertinent technology if it is chosen and measures of decision quality; Secondary outcomes include indices of metabolic control, quality of life and parent-adolescent relationships around diabetes management.

DETAILED DESCRIPTION:
Abstract (modified after achievement of Aims 1 and 2):

Treatment adherence in type 1 diabetes (T1D) tends to decline among adolescents, increasing risks of acute and chronic complications, excess health care use, poorer quality of life, and T1D-related family conflict. Poor adherence is associated with psychiatric and family dysfunction and often persists into early adulthood. Therapeutic advances such as continuous subcutaneous insulin infusion (CSII or "insulin pump") and continuous glucose monitoring (CGM) could improve metabolic control and quality of life.

But, teens often do not benefit fully from such advances. Many studies of adults show that patient-centered communication styles predict more favorable clinical outcomes. Shared medical decision making (SMDM) interventions have improved outcomes among adults with diabetes and other conditions. Research in pediatrics has also shown that patient-centered and family-centered communication styles predict favorable outcomes, but most of this research is in primary care and has not studied youth with chronic conditions. Since there have been no controlled trials of SMDM with chronically ill youths, we propose a randomized controlled trial of an SMDM intervention compared with Usual Clinical Practice (UCP). Qualitative interviews of youths and parents who have previously faced these decisions and reliance on expert consultants, pediatric endocrinologists and diabetes educators have preceded this trial and provided valued input for refining the planned intervention and adapting the structured SMDM format for pediatrics. Now, we will recruit and randomize 166 11-<17 year old youth with T1D who are candidates for CSII or CGM (and a parent/caregiver) at all Nemours sites. The SMDM intervention will be delivered via a web-based platform, facilitated by Diabetes Educators (DEs) at each site in a standardized, yet individually tailored format. SMDM will employ multimedia "decision aids" prepared with the award-winning Nemours Center for Children's Health Media and the "e-city interactive" web design firm in Philadelphia in accord with pertinent international standards. SMDM will also include individualized assistance from the DE in assuring that each youth's and parent's preferences, values and cultural beliefs are carefully addressed and communicated to the attending endocrinologist. After a baseline evaluation and randomization to SMDM or UCP, effects on the primary outcome (treatment adherence; device utilization) and secondary outcomes (glycemic control, treatment alliance, decision conflict and regret, treatment satisfaction, diabetes-related distress and self-efficacy) will be measured over 1 year. Mixed effects modeling will be the primary analytic technique for evaluating effects on primary/secondary outcomes, examining selected variables as moderators and mediators of treatment effects, and assessing whether such effects are comparable for the two medical decisions of interest. The results will verify whether SMDM in this context enhances treatment adherence, device use and parent/patient-reported outcomes in youth with T1D.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes for 1 year or more
* At least 2 diabetes clinic visits at the enrolling site in the prior year
* Considered by treating endocrinologist to be a candidate for insulin pump or continuous glucose monitor
* Intent to continue care at Nemours for 1 year
* Internet access at home, school, work or relative's home

Exclusion Criteria:

* Open case with child protection agency
* Unable to read and speak English

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 153 (Actual)
Dates: Start 2015-02; Primary Completion 2017-02-07 (Actual); Study Completion 2017-02-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tim Wysocki, PhD, Principal Investigator — Nemours Biomedical Research
Locations (1):
- Nemours Children's Clinic, Jacksonville, Florida, United States

REFERENCES:
- [Background] Wysocki T, Hirschfeld F, Miller L, Izenberg N, Dowshen SA, Taylor A, Milkes A, Shinseki MT, Bejarano C, Kozikowski C, Kowal K, Starr-Ashton P, Ross JL, Kummer M, Carakushansky M, Lyness D, Brinkman W, Pierce J, Fiks A, Christofferson J, Rafalko J, Lawson ML. Consideration of Insulin Pumps or Continuous Glucose Monitors by Adolescents With Type 1 Diabetes and Their Parents: Stakeholder Engagement in the Design of Web-Based Decision Aids. Diabetes Educ. 2016 Aug;42(4):395-407. doi: 10.1177/0145721716647492. Epub 2016 May 4. PMID 27150606

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred from 2015-2017 at all locations of Nemours Children's Health System (Wilmington, DE, Philadelphia, PA and Jacksonville, Orlando and Pensacola, FL. In 2017, the Barbara Davis Center for Childhood Diabetes in Denver was added as a performance site.
Pre-assignment Details: Of the 153 adolescent-parent dyads who provided consent/assent, 20 dyads did not complete all required baseline measures and were not randomized. 133 dyads were randomized to Usual Clinical Practice or Shared Decision Making.
Units Other Than Participants: Adolescent-Parent dyads
Groups:
- Usual Clinical Practice (UCP): UCP participants received the same clinical and educational management for candidates for insulin pump or continuous glucose monitoring that is received by similar patients who are not enrolled in this study. The respective endocrinology practices at the enrolling sites all strive to meet or exceed the current American Diabetes Association Standards for Clinical Practice in the management of type 1 diabetes in this population. Thorough patient education is the cornerstone of that care, especially regarding the incorporation of insulin pumps and continuous glucose monitors into the treatment regimen for a given patient.
  Usual Clinical Practice: Diabetes management and education related to insulin pump or continuous glucose monitor as currently practiced at the enrolling site.
- Shared Medical Decision Making (SMDM): Participants randomized to SMDM received all components of UCP supplemented with access to the decision aid website pertinent to the medical decision of interest (pump, CGM or both). Adolescents and parents received password-protected, secure access to the decision for their use until a decision was reached. The platform generated a summary report that the adolescent and parent could discuss with a diabetes nurse and then a visit with the treating endocrinologist was scheduled to conclude the SMDM intervention for that adolescent and parent.
  Shared Medical Decision Making: Access to and use of multimedia decision aid websites to facilitate adolescent and parent decision making about incorporating these devices into the diabetes management regimen.
Period: Overall Study
Arm/Group | Usual Clinical Practice (UCP) | Shared Medical Decision Making (SMDM)
Started | 67; 67 Adolescent-Parent dyads | 66; 66 Adolescent-Parent dyads
Completed | 62; 62 Adolescent-Parent dyads | 53; 53 Adolescent-Parent dyads
Not Completed | 5; 5 Adolescent-Parent dyads | 13; 13 Adolescent-Parent dyads
Not completed — Lost to Follow-up | 5 | 0
Not completed — 13SDM dyads did not access Decision Aids | 0 | 13

BASELINE CHARACTERISTICS:
Population: The population of interest consists of adolescents with type 1 diabetes and their parents who are considered by their attending diabetes care provider to be candidates for incorporation of either the insulin pump or continuous glucose monitoring into their diabetes treatment regimens.
Groups:
- Usual Clinical Practice (UCP): UCP participants received the same clinical and educational management for candidates for insulin pump or continuous glucose monitoring received by similar patients who were not enrolled in this study. The respective endocrinology practices at the enrolling sites all strive to meet or exceed the current American Diabetes Association Standards for Clinical Practice in the management of type 1 diabetes in this population. Thorough patient education is the cornerstone of that care, especially regarding the incorporation of insulin pumps and continuous glucose monitors into the treatment regimen for a given patient.
  Usual Clinical Practice: Diabetes management and education related to insulin pump or continuous glucose monitor as currently practiced at the enrolling site.
- Shared Medical Decision Making (SMDM): Participants randomized to SMDM received all components of UCP supplemented with access to the decision aid website pertinent to the medical decision of interest (pump or CGM). Adolescents and parents received password-protected, secure access to the decision for their use until a decision was reached. The platform then generated a summary report that the adolescent and parent could discuss with a diabetes nurse and then a visit with the treating endocrinologist was scheduled to conclude the SMDM intervention for that adolescent and parent.
  Shared Medical Decision Making: Access to and use of multimedia decision aid websites to facilitate adolescent and parent decision making about incorporating these devices into the diabetes management regimen.
- Total: Total of all reporting groups
Arm/Group | Usual Clinical Practice (UCP) | Shared Medical Decision Making (SMDM) | Total
Number analyzed (Participants) | 67 | 66 | 133
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 67 | 66 | 133
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.9 (2.0) | 13.5 (2.0) | 13.7 (1.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 34 | 65
  Male | 36 | 32 | 68
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 5 | 18
  Not Hispanic or Latino | 54 | 61 | 115
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 5 | 11
  White | 49 | 55 | 104
  More than one race | 5 | 3 | 8
  Unknown or Not Reported | 5 | 2 | 7
Region of Enrollment [Number; unit: participants]
  United States | 67 | 66 | 133
Hollingshead Four Factor Index of Social Status [Mean (Standard Deviation); unit: units on a scale] — The Hollingshead Index of Social Status provides an overall estimate of household socioeconomic status based on parents' categorizations of each parent's educational attainment and occupational category. Scores may range from 16 to 66, with higher scores indicative of higher educational attainment and occupational status.
  units on a scale | 45.7 (14.2) | 43.9 (13.1) | 44.9 (13.8)
Rapid Estimate of Adult/Adolescent Literacy in Medicine [Mean (Standard Deviation); unit: units on a scale] — This is a brief practical test of health literacy consisting of comprehension of health-related vocabulary terms. Higher scores indicate more proficient health literacy. Scores may range from 15 to 75.
  units on a scale | 62.9 (3.44) | 61.2 (4.93) | 62.1 (3.89)
Diabetes Numeracy Test [Mean (Standard Deviation); unit: units on a scale] — This is a brief practical assessment of one's health-related quantitative skills based on reading and comprehension of food labels and medication labels. Higher scores indicate stronger health numeracy skills. Scores may range from 0 to 15.
  units on a scale | 10.3 (2.48) | 11.0 (3.41) | 10.7 (2.99)
CGM/Insulin Pump Knowledge Test [Mean (Standard Deviation); unit: units on a scale] — These are brief tests of parent and adolescent knowledge of continuous glucose monitors and insulin pumps, respectively. Scores may range from 15-45 with higher scores reflecting greater knowledge of the diabetes device of interest.
  units on a scale | 36.7 (5.34) | 41.29 (5.09) | 39.1 (5.23)
Hemoglobin A1C [Mean (Standard Deviation); unit: percent] — HbA1c expressed as a percentage of hemoglobin molecules that are bound to glucose molecules. Higher values reflect increasingly high average blood glucose levels over the prior 2-3 months. Normal range is 4.5% to 6.5%.
  percent | 8.61 (1.29) | 8.53 (1.49) | 8.58 (1.41)

OUTCOME MEASURES:

1. Primary Outcome: Continuous Glucose Monitor Use Profile or Insulin Pump Use Profile
Description: Adolescent and Parent report regarding degree to which use of the device of interest has become an integral part of the adolescent's daily diabetes self management. Scores may range from 10 to 50, with higher scores reflecting more frequent and meticulous use of the diabetes device of interest.
Time Frame: Measure was collected at each study visit after the participant actually obtained a CGM or Insulin Pump
Population: The population of interest consists of adolescents with type 1 diabetes and their parents who are considered to be candidates for adoption of either the insulin pump or continuous glucose monitor as a component of their diabetes management regimens.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Usual Clinical Practice (UCP): UCP participants received the same clinical and educational management for candidates for insulin pump or continuous glucose monitoring that is received by similar patients who were not enrolled in this study. The respective endocrinology practices at the enrolling sites all strive to meet or exceed the current American Diabetes Association Standards for Clinical Practice in the management of type 1 diabetes in this population. Thorough patient education is the cornerstone of that care, especially regarding the incorporation of insulin pumps and continuous glucose monitors into the treatment regimen for a given patient.
  Usual Clinical Practice: Diabetes management and education related to insulin pump or continuous glucose monitor as currently practiced at the enrolling site.
- Shared Medical Decision Making (SMDM): Participants randomized to SMDM received all components of UCP supplemented with access to the decision aid website pertinent to the medical decision of interest (pump or CGM). Adolescents and parents received password-protected, secure access to the decision for their use until a decision is reached. The platform then generated a summary report that the adolescent and parent could discuss with a diabetes nurse and then a visit with the treating endocrinologist was scheduled to conclude the SMDM intervention for that adolescent and parent.
  Shared Medical Decision Making: Access to and use of multimedia decision aid websites to facilitate adolescent and parent decision making about incorporating these devices into the diabetes management regimen.
Arm/Group | Usual Clinical Practice (UCP) | Shared Medical Decision Making (SMDM)
Number analyzed (Participants) | 62 | 53
score on a scale
  Visit 2-Adolescents | 32.5 (4.3) | 34.2 (3.9)
  Visit 2-Parents | 40.1 (3.7) | 35.7 (5.1)
  Visit 3-Adolescents | 33.8 (4.7) | 33.7 (3.7)
  Visit Visit 3-Parents | 30.2 (3.1) | 35.1 (4.6)
  Visit 4-Adolescents | 33.7 (5.8) | 33.5 (4.8)
  Visit 4-Parents | 34.6 (4.3) | 32.1 (4.3)
  Visit 5-Adolescents | 33.3 (4.9) | 30.1 (4.7)
  Visit 5-Parents | 34.4 (5.6) | 33.3 (5.1)
Statistical Analysis 1: Comparison: Usual Clinical Practice (UCP) vs Shared Medical Decision Making (SMDM); Missing data treatment was done using multiple imputation methods when data were determined to be Missing Completely at Random or Missing at Random. Assumptions underlying each statistical test were evaluated before proceeding with specific analyses; Test type: Superiority; p < 0.39, Mixed Models Analysis — This is a computed p-value; For each outcome, a linear mixed effects model was fit; with the exception of the Knowledge test where a linear model was fit. Separate models were fit for Parents and adolescents except for HbA1C. The predictor variable is treatment group (SMDM vs. UCP). Covariates are gender, age, social economic status, and family structure as determined by (number of siblings and of caregivers in the home). A random intercept was fit for each subject across the longitudinal data. To accommodate missing values multiple imputation methodology was applied to the data, resulting in five imputed datasets. For each imputed dataset, a linear mixed effects model (or linear model for Knowledge Test) was fit; the resulting five models were pooled into a final model and summary statistics are presented. A two-sided Wald's t test determined significance of covariates. The significance level was 0.05. Appropriate model diagnostics were performed to assess model fit

2. Secondary Outcome: Glycated Hemoglobin (Hemoglobin A1C)
Description: Glycated hemoglobin (Hemoglobin A1C) expressed as the percentage of hemoglobin molecules that are bound to glucose. Normal range is approximately 4.5% to 6.5%, Higher values indicate a higher blood glucose concentration over the preceding 2-3 months.
Time Frame: Every 3 months for for 1 year
Population: Adolescents with type 1 diabetes and their parents who are considered by their attending diabetes care providers to be candidates for incorporation of the insulin pump or continuous glucose monitoring into their treatment regimens.
Measure: Mean (Standard Deviation); unit: percentage (HbA1c)
Arm/Group | Usual Clinical Practice (UCP) | Shared Medical Decision Making (SMDM)
Number analyzed (Participants) | 62 | 53
percentage (HbA1c)
  Visit 1 | 8.61 (1.29) | 8.53 (1.49)
  Visit 2 | 8.54 (1.30) | 8.24 (1.25)
  Visit 3 | 8.80 (1.48) | 8.55 (1.48)
  Visit 4 | 9.24 (2.03) | 8.59 (1.29)
  Visit 5 | 8.69 (1.43) | 8.83 (1.95)
Statistical Analysis 1: Comparison: Usual Clinical Practice (UCP) vs Shared Medical Decision Making (SMDM); Test type: Superiority; p > 0.05, Mixed Models Analysis — Computed p-value exceeded the .05 level of significance; [other analysis details as in outcome 1, analysis 1]

3. Secondary Outcome: Decision Regret Scale
Description: Questionnaire measuring decision making regret. Reflecting on a specific decision (accept or decline opportunity to use CGM or insulin pump), higher score reflect a greater degree of regret regarding the decision that was made. Scores may range from 5 to 20.
Time Frame: Obtained at Visits 3 and 5 only
Population: Adolescents with type 1 diabetes and their parents who are considered by their diabetes care providers to be candidates for incorporation of insulin pump or CGM into their treatment regimens.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Clinical Practice (UCP) | Shared Medical Decision Making (SMDM)
Number analyzed (Participants) | 62 | 53
score on a scale
  Visit 3 | 9.14 (3.70) | 9.85 (4.07)
  Visit 5 | 8.69 (3.11) | 8.53 (3.08)
Statistical Analysis 1: Comparison: Usual Clinical Practice (UCP) vs Shared Medical Decision Making (SMDM); See description of analysis below; Test type: Superiority; p > 0.05, Mixed Models Analysis — This is a computed p-value; [other analysis details as in outcome 1, analysis 1]

4. Secondary Outcome: Knowledge of Insulin Pump or Continuous Glucose Monitor
Description: Brief test of parent and adolescent knowledge about the pertinent device and its use. Higher scores reflect more precise knowledge about the diabetes device of interest. Scores may range from 1 to 5.
Time Frame: Baseline and 3 months later
Population: Adolescents with T1D and their parents considering adoption of CSII or CGM.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Clinical Practice (UCP) | Shared Medical Decision Making (SMDM)
Number analyzed (Participants) | 62 | 53
score on a scale
  Visit 1 | 2.86 (1.18) | 2.76 (1.21)
  Visit 2 | 3.14 (1.14) | 3.40 (1.11)
Statistical Analysis 1: Comparison: Usual Clinical Practice (UCP) vs Shared Medical Decision Making (SMDM); Test type: Superiority; p > 0.05, ANCOVA — Computed p-value; Difference in post-test scores with baseline Knowledge test score as the covariate

5. Secondary Outcome: Diabetes Self Management Profile Self Report Form
Description: Composite measure of diabetes treatment adherence consisting of combined scores based on reports of parents and adolescents. Higher scores reflect more meticulous adherence to recommended diabetes self management behaviors. Scores may range from 0 to 86.
Time Frame: Visits 1, 3 and 5
Population: Adolescents with T1D and parents considering adoption of CSII or CGM.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Clinical Practice (UCP) | Shared Medical Decision Making (SMDM)
Number analyzed (Participants) | 62 | 53
score on a scale
  Visit 1 | 55.03 (10.66) | 56.19 (10.03)
  Visit 3 | 55.91 (10.83) | 56.25 (11.17)
  Visit 5 | 56.08 (11.98) | 54.14 (12.27)

6. Secondary Outcome: SURE Test
Description: 4-item questionnaire that measures patients' confidence in a health care decision that has been made. Scores may range from 0-4 with higher scores reflecting greater confidence in the decision made regarding insulin pump or CGM.
Time Frame: Measured at Follow-up Visits 3 and 5 only
Population: Adolescents with T1D and parents considering adoption of CSII or CGM.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Clinical Practice (UCP) | Shared Medical Decision Making (SMDM)
Number analyzed (Participants) | 62 | 53
score on a scale
  Visit 3 | 3.43 (0.74) | 3.74 (0.50)
  Visit 5 | 3.70 (0.56) | 3.73 (0.46)
Statistical Analysis 1: Comparison: Usual Clinical Practice (UCP) vs Shared Medical Decision Making (SMDM); Test type: Superiority — See analysis description below; p > 0.05, ANOVA — Computed p-value; [other analysis details as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Each participant was monitored for study-related and unanticipated adverse events for 1 year during study participation.
Description: This trial was educational in nature and the intervention did nothing more than to expose adolescents and parents to the best available information pertinent to deciding whether or not to adopt an insulin pump or continuous glucose monitor as a component of the adolescent's diabetes regimen. The trial was considered by the IRB to pose no greater than minimal risk to participants.
Groups:
- Usual Clinical Practice (UCP): UCP participants received the same clinical and educational management for candidates for insulin pump or continuous glucose monitoring that was received by similar patients who were not enrolled in this study. The respective endocrinology practices at the enrolling sites all strive to meet or exceed the current American Diabetes Association Standards for Clinical Practice in the management of type 1 diabetes in this population. Thorough patient education is the cornerstone of that care, especially regarding the incorporation of insulin pumps and continuous glucose monitors into the treatment regimen for a given patient.
  Usual Clinical Practice: Diabetes management and education related to insulin pump or continuous glucose monitor as currently practiced at the enrolling site.
Arm/Group | Usual Clinical Practice (UCP) | Shared Medical Decision Making (SMDM)
All-Cause Mortality (participants affected / at risk) | 0/67 | 0/66
Serious Adverse Events (participants affected / at risk) | 0/67 | 0/67
Other Adverse Events (participants affected / at risk) | 0/67 | 0/66

LIMITATIONS AND CAVEATS:
A small percentage of all adolescents entering the study actually proceeded to acquire an insulin pump or continuous glucose monitor during the study period, impeding analyses of the effects of the SDM intervention on scores on the CGM Use Profile

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-03-28): https://cdn.clinicaltrials.gov/large-docs/56/NCT02496156/Prot_SAP_000.pdf
  • Informed Consent Form (2016-11-07): https://cdn.clinicaltrials.gov/large-docs/56/NCT02496156/ICF_001.pdf